CLINICAL TRIAL: NCT01730534
Title: Dapagliflozin Effect on Cardiovascular Events A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effect of Dapagliflozin 10 mg Once Daily on the Incidence of Cardiovascular Death, Myocardial Infarction or Ischemic Stroke in Patients With Type 2 Diabetes
Brief Title: Multicenter Trial to Evaluate the Effect of Dapagliflozin on the Incidence of Cardiovascular Events
Acronym: DECLARE-TIMI58
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry); The TIMI Study Group (Other); Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1693C00001
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; High Risk for Cardiovascular Event
Keywords: Phase IIIb; T2DM; cardiovascular events
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin + standard of care therapy for Type 2 Diabetes and for co-morbidities and cardiovascular risk factors
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo (Placebo Comparator): Placebo + standard of care therapy for Type 2 Diabetes and for co-morbidities and cardiovascular risk factors
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Oral dose (od)
  Arms: Dapagliflozin
Drug: Placebo tablet — Oral dose (od)
  Arms: Placebo

SUMMARY:
This study is being carried out to determine the effect of dapagliflozin on cardiovacular outcomes when added to current background therapy in patients with type 2 diabetes with either established cardiovacular disease or cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female or male aged ≥40 years
* Diagnosed with Type 2 Diabetes
* High Risk for Cardiovascular events

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus History of bladder cancer or history of radiation therapy to the lower abdomen or pelvis at any time
* Chronic cystitis and/or recurrent urinary tract infections
* Pregnant or breast-feeding patients

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17190 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Langkilde, MD, Study Director — AstraZeneca Sweden; Marc S Sabatine, MD, MPH, Study Chair — TIMI Study Group, Boston, MA, USA; Itamar Raz, MD, Principal Investigator — Hadassah Medical Organization; Stephen D Wiviott, MD, Principal Investigator — TIMI Study Group, MA, USA
Locations (641):
- United States (205):
  - Research Site, Alexander City, Alabama
  - Research Site, Athens, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Alhambra, California
  - Research Site, Bakersfield, California
  - Research Site, Greenbrae, California
  - Research Site, Huntington Park, California
  - Research Site, La Mesa, California
  - Research Site, Lomita, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, San Diego, California
  - Research Site, San Marino, California
  - Research Site, San Ramon, California
  - Research Site, Torrance, California
  - Research Site, Ventura, California
  - Research Site, Vista, California
  - Research Site, Fort Collins, Colorado
  - Research Site, Golden, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Bristol, Connecticut
  - Research Site, Norwalk, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Seaford, Delaware
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bradenton, Florida
  - Research Site, Chiefland, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Green Cove Springs, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Ocala, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Spring Hill, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Stuart, Florida
  - Research Site, Tampa, Florida
  - Research Site, Trinity, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Wellington, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Calhoun, Georgia
  - Research Site, Cumming, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Arlington Heights, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Rock Island, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Avon, Indiana
  - Research Site, Bloomington, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Greenfield, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Newburgh, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Hammond, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Biddeford, Maine
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Beltsville, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Methuen, Massachusetts
  - Research Site, Natick, Massachusetts
  - Research Site, Alpena, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Grand Blanc, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Eagan, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Lee's Summit, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Great Falls, Montana
  - Research Site, Kalispell, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Reno, Nevada
  - Research Site, Edison, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Northport, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Southampton, New York
  - Research Site, Stony Brook, New York
  - Research Site, Westfield, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Canal Fulton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Delaware, Ohio
  - Research Site, Elyria, Ohio
  - Research Site, Parma Hts., Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Altoona, Pennsylvania
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Indiana, Pennsylvania
  - Research Site, Johnstown, Pennsylvania
  - Research Site, Kittanning, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Tyrone, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Katy, Texas
  - Research Site, Kingwood, Texas
  - Research Site, McAllen, Texas
  - Research Site, Midland, Texas
  - Research Site, Odessa, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Tyler, Texas
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Bennington, Vermont
  - Research Site, Burke, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Burien, Washington
  - Research Site, Puyallup, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Wausau, Wisconsin
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Lanús
  - Research Site, Mar del Plata
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, San Nicolás
  - Research Site, Santa Fe
- Australia (16):
  - Research Site, Adelaide - Oaklands Park
  - Research Site, Ashford
  - Research Site, Box Hill
  - Research Site, Camperdown
  - Research Site, Darlinghurst
  - Research Site, Fullarton
  - Research Site, Garran
  - Research Site, Geelong
  - Research Site, Heidelberg West
  - Research Site, Herston
  - Research Site, Joondalup
  - Research Site, Maroubra
  - Research Site, Melbourne
  - Research Site, Milton
  - Research Site, Murdoch
  - Research Site, Wollongong
- Belgium (14):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Bonheiden
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Merksem
  - Research Site, Roeselare
  - Research Site, Tienen
  - Research Site, Turnhout
- Brazil (9):
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Marília
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
  - Research Site, São José dos Campos
  - Research Site, São Paulo
- Bulgaria (19):
  - Research Site, Blagoevgrad
  - Research Site, Botevgrad
  - Research Site, Dimitrovgrad
  - Research Site, Dupnitsa
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Kyustendil
  - Research Site, Lukovit
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Yambol
- Canada (33):
  - Research Site, Calgary, Alberta
  - Research Site, New Westminster, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney Mines, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Concord, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Georges, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Laval
- China (10):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
- Czechia (24):
  - Research Site, Beroun
  - Research Site, Brno
  - Research Site, Cheb
  - Research Site, Chomutov
  - Research Site, Chrudim III
  - Research Site, Hodonín
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Jílové u Prahy
  - Research Site, Kroměříž
  - Research Site, Ostrava - Belsky Les
  - Research Site, Ostrava - Dubina
  - Research Site, Ostrava-Kunčice
  - Research Site, Ostrava-Moravska
  - Research Site, Pilsen
  - Research Site, Plzen - Severni Predmesti
  - Research Site, Prague
  - Research Site, Přelouč
  - Research Site, Rakovník
  - Research Site, Slaný
  - Research Site, Teplice
  - Research Site, Uherské Hradiště
  - Research Site, Ústí nad Labem
  - Research Site, Zlín
- France (9):
  - Research Site, Angers
  - Research Site, Corbeil-Essonnes
  - Research Site, Dijon
  - Research Site, La Rochelle
  - Research Site, Le Creusot
  - Research Site, Nantes
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Toulouse
- Germany (12):
  - Research Site, Aschaffenburg
  - Research Site, Bad Mergentheim
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dippoldiswalde
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Villingen-Schwenningen
- Hong Kong (3):
  - Research Site, Causeway Bay
  - Research Site, Hong Kong
  - Research Site, Tai Po
- Hungary (23):
  - Research Site, Ács
  - Research Site, Balatonfüred
  - Research Site, Ballasagyarmat
  - Research Site, Berettyóújfalu
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Csongrád
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Esztergom
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Kistarcsa
  - Research Site, Komárom
  - Research Site, Mórahalom
  - Research Site, Nyíregyháza
  - Research Site, Polgár
  - Research Site, Sopron
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Tát
  - Research Site, Zalaegerszeg
- India (4):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Pune
  - Research Site, Vellore
- Israel (10):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Bnei Barak
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikva
- Italy (12):
  - Research Site, Bergamo
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Negrar - VR
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Rozzano
  - Research Site, S Maria Capua Vetere
  - Research Site, Sessa Aurunca
  - Research Site, Verona
- Japan (11):
  - Research Site, Bunkyō City
  - Research Site, Daito-shi
  - Research Site, Kasuga-shi
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Matsubara-shi
  - Research Site, Saga
  - Research Site, Ube-shi
  - Research Site, Uji-shi
  - Research Site, Yakushi
  - Research Site, Yokohama
- Mexico (16):
  - Research Site, Acapulco
  - Research Site, Culiacán
  - Research Site, Del. Cuauhtemoc
  - Research Site, Distrito Federal
  - Research Site, Guadalajara
  - Research Site, Meridas
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Pachuca
  - Research Site, Querétaro
  - Research Site, San Luis Potosí City
  - Research Site, Tijuana
  - Research Site, Veracruz
  - Research Site, Xalapa
  - Research Site, Zapopan
  - Research Site, Zapopan, Jalisco
- Netherlands (22):
  - Research Site, Alkmaar
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Delft
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Hardenberg
  - Research Site, Heerlen
  - Research Site, Hoogeveen
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Sliedrecht
  - Research Site, Sneek
  - Research Site, The Hague
  - Research Site, Utrecht
  - Research Site, Venlo
  - Research Site, Zutphen
- Philippines (13):
  - Research Site, Bacolod
  - Research Site, Cebu City
  - Research Site, Dasmariñas
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Makati City
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasay
  - Research Site, Pasig
  - Research Site, Quezon City
  - Research Site, Tanauan
- Poland (27):
  - Research Site, Biała Rawska
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Giżycko
  - Research Site, Katowice
  - Research Site, Koluszki
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Lublin
  - Research Site, Mrągowo
  - Research Site, Nakło nad Notecią
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Skierniewice
  - Research Site, Sobótka
  - Research Site, Sokółka
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Węgrów
  - Research Site, Wierzchosławice
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zabrze
  - Research Site, Łęczna
- Romania (12):
  - Research Site, Bacau
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Galati
  - Research Site, Iași
  - Research Site, Ploieşti
  - Research Site, Sibiu
  - Research Site, Târgu Mures
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
  - Research Site, Zalău
- Russia (17):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
- Slovakia (19):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Námestovo
  - Research Site, Nové Zámky
  - Research Site, Piešťany
  - Research Site, Poprad
  - Research Site, Považská Bystrica
  - Research Site, Prievidza
  - Research Site, Rimavská Sobota
  - Research Site, Sabinov
  - Research Site, Šaľa
  - Research Site, Trebišov
  - Research Site, Trenčín
  - Research Site, Vrútky
  - Research Site, Žilina
- South Africa (14):
  - Research Site, Alberton
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Diepkloof, Soweto
  - Research Site, Durban
  - Research Site, Goodwood
  - Research Site, Houghton Estate
  - Research Site, Muckleneuk
  - Research Site, Parktown
  - Research Site, Parktown West
  - Research Site, Phoenix
  - Research Site, Somerset West
  - Research Site, Verulam
  - Research Site, Worcester
- South Korea (13):
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Jeonju-si, Jeollabuk-do
  - Research Site, Junggu
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
- Spain (8):
  - Research Site, Almería
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Sant Joan Despí
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- Sweden (13):
  - Research Site, Borås
  - Research Site, Eksjö
  - Research Site, Finspång
  - Research Site, Gothenburg
  - Research Site, Järfälla
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Östersund
  - Research Site, Rättvik
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Vällingby
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (9):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Muang
  - Research Site, Nakhon Ratchasima
  - Research Site, Pathum Thani
  - Research Site, Phisanulok
  - Research Site, Rajthevi
  - Research Site, Ratchaburi
  - Research Site, Ratchathewi
- Turkey (Türkiye) (3):
  - Research Site, Antalya
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (9):
  - Research Site, Dnipro
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Vinnytsia
  - Research Site, Vynnitsa
  - Research Site, Zaporizhzhya
- United Kingdom (14):
  - Research Site, Addlestone
  - Research Site, Aylesbury
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Canterbury
  - Research Site, Corsham
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Irvine
  - Research Site, Leicester
  - Research Site, Mortimer Reading
  - Research Site, Sheffield
  - Research Site, Whitstable
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Haller PM, Wiviott SD, Berg DD, Jarolim P, Goodrich EL, Bhatt DL, Gause-Nilsson I, Leiter LA, McGuire DK, Wilding JPH, Raz I, Sabatine MS, Morrow DA. Galectin-3 and kidney function in type 2 diabetes treated with dapagliflozin: Analysis from DECLARE-TIMI 58. ESC Heart Fail. 2025 Dec;12(6):3981-3986. doi: 10.1002/ehf2.15415. Epub 2025 Sep 15. PMID 40952180
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Schechter M, Wiviott SD, Raz I, Goodrich EL, Rozenberg A, Yanuv I, Murphy SA, Zelniker TA, Fredriksson M, Johansson PA, Leiter LA, Bhatt DL, McGuire DK, Wilding JPH, Gause-Nilsson IAM, Cahn A, Langkilde AM, Sabatine MS, Mosenzon O. Effects of dapagliflozin on hospitalisations in people with type 2 diabetes: post-hoc analyses of the DECLARE-TIMI 58 trial. Lancet Diabetes Endocrinol. 2023 Apr;11(4):233-241. doi: 10.1016/S2213-8587(23)00009-8. Epub 2023 Mar 3. PMID 36878239
- [Derived] Zelniker TA, Wiviott SD, Mosenzon O, Goodrich EL, Jarolim P, Cahn A, Bhatt DL, Leiter LA, McGuire DK, Wilding J, Averkov O, Budaj A, Parkhomenko A, Ray KK, Gause-Nilsson I, Langkilde AM, Fredriksson M, Raz I, Sabatine MS, Morrow DA. Association of Cardiac Biomarkers With Major Adverse Cardiovascular Events in High-risk Patients With Diabetes: A Secondary Analysis of the DECLARE-TIMI 58 Trial. JAMA Cardiol. 2023 May 1;8(5):503-509. doi: 10.1001/jamacardio.2023.0019. PMID 36857035
- [Derived] Mosenzon O, Raz I, Wiviott SD, Schechter M, Goodrich EL, Yanuv I, Rozenberg A, Murphy SA, Zelniker TA, Langkilde AM, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Wilding JPH, McGuire DK, Bhatt DL, Leiter LA, Cahn A, Dwyer JP, Heerspink HJL, Sabatine MS. Dapagliflozin and Prevention of Kidney Disease Among Patients With Type 2 Diabetes: Post Hoc Analyses From the DECLARE-TIMI 58 Trial. Diabetes Care. 2022 Oct 1;45(10):2350-2359. doi: 10.2337/dc22-0382. PMID 35997319
- [Derived] Oyama K, Raz I, Cahn A, Goodrich EL, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Gause-Nilsson IAM, Mosenzon O, Sabatine MS, Wiviott SD. Efficacy and Safety of Dapagliflozin According to Background Use of Cardiovascular Medications in Patients With Type 2 Diabetes: A Prespecified Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2022 Sep 1;7(9):914-923. doi: 10.1001/jamacardio.2022.2006. PMID 35857296
- [Derived] Furtado RHM, Raz I, Goodrich EL, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Aylward P, Dalby AJ, Dellborg M, Dimulescu D, Nicolau JC, Oude Ophuis AJM, Cahn A, Mosenzon O, Gause-Nilsson I, Langkilde AM, Sabatine MS, Wiviott SD. Efficacy and Safety of Dapagliflozin in Type 2 Diabetes According to Baseline Blood Pressure: Observations From DECLARE-TIMI 58 Trial. Circulation. 2022 May 24;145(21):1581-1591. doi: 10.1161/CIRCULATIONAHA.121.058103. Epub 2022 May 5. PMID 35510542
- [Derived] Cahn A, Wiviott SD, Mosenzon O, Goodrich EL, Murphy SA, Yanuv I, Rozenberg A, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Gause-Nilsson IAM, Langkilde AM, Sabatine MS, Raz I. Association of Baseline HbA1c With Cardiovascular and Renal Outcomes: Analyses From DECLARE-TIMI 58. Diabetes Care. 2022 Apr 1;45(4):938-946. doi: 10.2337/dc21-1744. PMID 35015847
- [Derived] Oyama K, Raz I, Cahn A, Kuder J, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Park KS, Goudev A, Diaz R, Spinar J, Gause-Nilsson IAM, Mosenzon O, Sabatine MS, Wiviott SD. Obesity and effects of dapagliflozin on cardiovascular and renal outcomes in patients with type 2 diabetes mellitus in the DECLARE-TIMI 58 trial. Eur Heart J. 2022 Aug 14;43(31):2958-2967. doi: 10.1093/eurheartj/ehab530. PMID 34427295
- [Derived] Mosenzon O, Wiviott SD, Heerspink HJL, Dwyer JP, Cahn A, Goodrich EL, Rozenberg A, Schechter M, Yanuv I, Murphy SA, Zelniker TA, Gause-Nilsson IAM, Langkilde AM, Fredriksson M, Johansson PA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Sabatine MS, Raz I. The Effect of Dapagliflozin on Albuminuria in DECLARE-TIMI 58. Diabetes Care. 2021 Aug;44(8):1805-1815. doi: 10.2337/dc21-0076. Epub 2021 Jul 7. PMID 34233928
- [Derived] Cherney DZI, Dagogo-Jack S, McGuire DK, Cosentino F, Pratley R, Shih WJ, Frederich R, Maldonado M, Liu J, Wang S, Cannon CP; VERTIS CV Investigators. Kidney outcomes using a sustained >/=40% decline in eGFR: A meta-analysis of SGLT2 inhibitor trials. Clin Cardiol. 2021 Aug;44(8):1139-1143. doi: 10.1002/clc.23665. Epub 2021 Jun 15. PMID 34129237
- [Derived] Zelniker TA, Raz I, Mosenzon O, Dwyer JP, Heerspink HHJL, Cahn A, Goodrich EL, Im K, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Gause-Nilsson I, Langkilde AM, Sabatine MS, Wiviott SD. Effect of Dapagliflozin on Cardiovascular Outcomes According to Baseline Kidney Function and Albuminuria Status in Patients With Type 2 Diabetes: A Prespecified Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2021 Jul 1;6(7):801-810. doi: 10.1001/jamacardio.2021.0660. PMID 33851953
- [Derived] Cahn A, Raz I, Leiter LA, Mosenzon O, Murphy SA, Goodrich EL, Yanuv I, Rozenberg A, Bhatt DL, McGuire DK, Wilding JPH, Gause-Nilsson IAM, Langkilde AM, Sabatine MS, Wiviott SD. Cardiovascular, Renal, and Metabolic Outcomes of Dapagliflozin Versus Placebo in a Primary Cardiovascular Prevention Cohort: Analyses From DECLARE-TIMI 58. Diabetes Care. 2021 May;44(5):1159-1167. doi: 10.2337/dc20-2492. Epub 2021 Mar 2. PMID 33653824
- [Derived] O'Donoghue ML, Kato ET, Mosenzon O, Murphy SA, Cahn A, Herrera M, Tankova T, Smahelova A, Merlini P, Gause-Nilsson I, Langkilde AM, McGuire DK, Wilding JPH, Leiter LA, Bhatt DL, Raz I, Sabatine MS, Wiviott SD. The efficacy and safety of dapagliflozin in women and men with type 2 diabetes mellitus. Diabetologia. 2021 Jun;64(6):1226-1234. doi: 10.1007/s00125-021-05399-2. Epub 2021 Feb 20. PMID 33611623
- [Derived] Bonaca MP, Wiviott SD, Zelniker TA, Mosenzon O, Bhatt DL, Leiter LA, McGuire DK, Goodrich EL, De Mendonca Furtado RH, Wilding JPH, Cahn A, Gause-Nilsson IAM, Johanson P, Fredriksson M, Johansson PA, Langkilde AM, Raz I, Sabatine MS. Dapagliflozin and Cardiac, Kidney, and Limb Outcomes in Patients With and Without Peripheral Artery Disease in DECLARE-TIMI 58. Circulation. 2020 Aug 25;142(8):734-747. doi: 10.1161/CIRCULATIONAHA.119.044775. Epub 2020 Aug 3. PMID 32795086
- [Derived] Zelniker TA, Bonaca MP, Furtado RHM, Mosenzon O, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Budaj A, Kiss RG, Padilla F, Gause-Nilsson I, Langkilde AM, Raz I, Sabatine MS, Wiviott SD. Effect of Dapagliflozin on Atrial Fibrillation in Patients With Type 2 Diabetes Mellitus: Insights From the DECLARE-TIMI 58 Trial. Circulation. 2020 Apr 14;141(15):1227-1234. doi: 10.1161/CIRCULATIONAHA.119.044183. Epub 2020 Jan 27. PMID 31983236
- [Derived] Cahn A, Mosenzon O, Wiviott SD, Rozenberg A, Yanuv I, Goodrich EL, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS, Raz I. Efficacy and Safety of Dapagliflozin in the Elderly: Analysis From the DECLARE-TIMI 58 Study. Diabetes Care. 2020 Feb;43(2):468-475. doi: 10.2337/dc19-1476. Epub 2019 Dec 16. PMID 31843945
- [Derived] Berg DD, Wiviott SD, Scirica BM, Gurmu Y, Mosenzon O, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Johanson P, Johansson PA, Langkilde AM, Raz I, Braunwald E, Sabatine MS. Heart Failure Risk Stratification and Efficacy of Sodium-Glucose Cotransporter-2 Inhibitors in Patients With Type 2 Diabetes Mellitus. Circulation. 2019 Nov 5;140(19):1569-1577. doi: 10.1161/CIRCULATIONAHA.119.042685. Epub 2019 Aug 31. PMID 31474116
- [Derived] Mosenzon O, Wiviott SD, Cahn A, Rozenberg A, Yanuv I, Goodrich EL, Murphy SA, Heerspink HJL, Zelniker TA, Dwyer JP, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Kato ET, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS, Raz I. Effects of dapagliflozin on development and progression of kidney disease in patients with type 2 diabetes: an analysis from the DECLARE-TIMI 58 randomised trial. Lancet Diabetes Endocrinol. 2019 Aug;7(8):606-617. doi: 10.1016/S2213-8587(19)30180-9. Epub 2019 Jun 10. PMID 31196815
- [Derived] Furtado RHM, Bonaca MP, Raz I, Zelniker TA, Mosenzon O, Cahn A, Kuder J, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Nicolau JC, Gause-Nilsson IAM, Fredriksson M, Langkilde AM, Sabatine MS, Wiviott SD. Dapagliflozin and Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus and Previous Myocardial Infarction. Circulation. 2019 May 28;139(22):2516-2527. doi: 10.1161/CIRCULATIONAHA.119.039996. Epub 2019 Mar 18. PMID 30882239
- [Derived] Kato ET, Silverman MG, Mosenzon O, Zelniker TA, Cahn A, Furtado RHM, Kuder J, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Bonaca MP, Ruff CT, Desai AS, Goto S, Johansson PA, Gause-Nilsson I, Johanson P, Langkilde AM, Raz I, Sabatine MS, Wiviott SD. Effect of Dapagliflozin on Heart Failure and Mortality in Type 2 Diabetes Mellitus. Circulation. 2019 May 28;139(22):2528-2536. doi: 10.1161/CIRCULATIONAHA.119.040130. Epub 2019 Mar 18. PMID 30882238
- [Derived] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Derived] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Bansilal S, Bhatt DL, Leiter LA, McGuire DK, Wilding JP, Gause-Nilsson IA, Langkilde AM, Johansson PA, Sabatine MS. The design and rationale for the Dapagliflozin Effect on Cardiovascular Events (DECLARE)-TIMI 58 Trial. Am Heart J. 2018 Jun;200:83-89. doi: 10.1016/j.ahj.2018.01.012. Epub 2018 Feb 7. PMID 29898853
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Eligibility varies among the 4 sodium-glucose cotransporter-2 inhibitor cardiovascular outcomes trials: implications for the general type 2 diabetes US population. Am J Manag Care. 2018 Apr;24(8 Suppl):S138-S145. PMID 29693360
- [Derived] Bloch MJ. Blood pressure effects of SGLT2 inhibitors make them an attractive option in diabetic patients with hypertension. J Am Soc Hypertens. 2016 Mar;10(3):186-7. doi: 10.1016/j.jash.2016.01.001. No abstract available. PMID 27408945
- [Derived] Leiter LA, Cefalu WT, de Bruin TW, Xu J, Parikh S, Johnsson E, Gause-Nilsson I. Long-term maintenance of efficacy of dapagliflozin in patients with type 2 diabetes mellitus and cardiovascular disease. Diabetes Obes Metab. 2016 Aug;18(8):766-74. doi: 10.1111/dom.12666. Epub 2016 May 12. PMID 27009868
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1693C00001&attachmentIdentifier=9c285ea0-c985-475c-9454-693ef18bed8c&fileName=DECLARE_TIMI_58_D1693C00001-revised-csp_5_Redacted_version.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1693C00001&attachmentIdentifier=0d14dc43-84c6-4ae3-a27d-b04c4a7b32a7&fileName=DECLARE_TIMI_58_Trial_D1693C00001_Statistical_Analysis_Plan_Redacted_version.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapa 10 mg: Dapagliflozin 10 mg tablets administered orally once daily
- Placebo: Matching placebo for dapagliflozin 10 mg administered orally once daily
Period: Overall Study
Arm/Group | Dapa 10 mg | Placebo
Started | 8582 | 8578
Completed | 8473 | 8433
Not Completed | 109 | 145
Not completed — Withdrawal by Subject | 97 | 127
Not completed — Lost to Follow-up | 12 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapa 10 mg | Placebo | Total
Number analyzed (Participants) | 8582 | 8578 | 17160
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.8) | 64.0 (6.8) | 63.9 (6.8)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 4631 | 4622 | 9253
  >=65 years | 3951 | 3956 | 7907
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 8044 | 8020 | 16064
  >=75 years | 538 | 558 | 1096
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3171 | 3251 | 6422
  Male | 5411 | 5327 | 10738
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1298 | 1270 | 2568
  Not Hispanic or Latino | 7284 | 7308 | 14592
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6843 | 6810 | 13653
  Black or African American | 295 | 308 | 603
  Asian | 1148 | 1155 | 2303
  American Indian or Alaska Native | 52 | 52 | 104
  Native Hawaiian or other Pacific Islander | 9 | 13 | 22
  Other | 235 | 240 | 475
Baseline CV risk category [Count of Participants; unit: Participants]
  Established CV disease | 3474 | 3500 | 6974
  Multiple risk factors for CV events | 5108 | 5078 | 10186

OUTCOME MEASURES:

1. Primary Outcome: Subjects Included in the Composite Endpoint of CV Death, MI or Ischemic Stroke
Description: Safety and co-primary efficacy
Time Frame: up to 5.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 8582 | 8578
Participants
  Number of patients with an event | 756 | 803
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Test type: Superiority; p = 0.172, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI [0.84 to 1.03]

2. Primary Outcome: Subjects Included in the Composite Endpoint of CV Death or Hospitalization Due to Heart Failure.
Description: Co-primary efficacy
Time Frame: up to 5.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 8582 | 8578
Participants
  Number of patients with an event | 417 | 496
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Test type: Superiority; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI [0.73 to 0.95]

3. Secondary Outcome: Subjects Included in the Renal Composite Endpoint: Confirmed Sustained ≥40% Decrease in eGFR to eGFR <60 ml/Min/1.73m2 and/or ESRD and/or Renal or CV Death.
Description: Secondary
Time Frame: up to 5.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 8582 | 8578
Participants
  Number of patients with an event | 370 | 480
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI [0.67 to 0.87]

4. Secondary Outcome: Subjects Included in the Endpoint of All-cause Mortality.
Description: Secondary
Time Frame: up to 5.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 8582 | 8578
Participants
  Number of patients with an event | 529 | 570
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Test type: Superiority; p = 0.198, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI [0.82 to 1.04]

ADVERSE EVENTS:
Time Frame: up to 5.2 years
Description: All-Cause Mortality was assessed for all participants. Serious and Other Adverse Events were only assessed for the Safety Analysis Population, which included participants that received at least one dose of study drug and who have data observed at any time after first randomized dose until the end of the study.
Groups:
- Dapa 10 mg; Placebo: Description (Arm-group)
Arm/Group | Dapa 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 529/8582 | 570/8578
Serious Adverse Events (participants affected / at risk) | 3205/8574 | 3418/8569
Other Adverse Events (participants affected / at risk) | 268/8574 | 342/8569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10 mg (N=8574) | Placebo (N=8569)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 20 (20) | 28 (30)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Elephantiasis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 12 (14) | 18 (18)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Plasmacytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic cyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute cardiac event (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 17 (22) | 31 (33)
Acute left ventricular failure (Cardiac disorders) | 16 (22) | 17 (23)
Acute myocardial infarction (Cardiac disorders) | 265 (293) | 233 (264)
Adams-stokes syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 154 (178) | 159 (175)
Angina unstable (Cardiac disorders) | 271 (349) | 269 (332)
Aortic valve calcification (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve disease (Cardiac disorders) | 3 (3) | 2 (2)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 10 (10) | 2 (2)
Arrhythmia (Cardiac disorders) | 5 (5) | 6 (6)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3) | 16 (21)
Atrial fibrillation (Cardiac disorders) | 117 (138) | 139 (177)
Atrial flutter (Cardiac disorders) | 21 (25) | 34 (44)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block (Cardiac disorders) | 2 (2) | 7 (7)
Atrioventricular block complete (Cardiac disorders) | 19 (19) | 14 (14)
Atrioventricular block second degree (Cardiac disorders) | 10 (10) | 7 (7)
Bifascicular block (Cardiac disorders) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 16 (17) | 21 (22)
Bundle branch block left (Cardiac disorders) | 0 (0) | 2 (2)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 33 (34) | 31 (32)
Cardiac asthma (Cardiac disorders) | 1 (1) | 5 (8)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 147 (199) | 188 (252)
Cardiac failure acute (Cardiac disorders) | 22 (25) | 31 (39)
Cardiac failure chronic (Cardiac disorders) | 12 (14) | 20 (23)
Cardiac failure congestive (Cardiac disorders) | 121 (177) | 147 (205)
Cardiac tamponade (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 5 (5)
Cardio-respiratory arrest (Cardiac disorders) | 12 (12) | 11 (11)
Cardiogenic shock (Cardiac disorders) | 19 (19) | 13 (16)
Cardiomegaly (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 7 (8) | 8 (8)
Cardiomyopathy acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 7 (7)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 3 (3)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 106 (113) | 84 (87)
Coronary artery occlusion (Cardiac disorders) | 9 (9) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 12 (13) | 22 (23)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Coronary ostial stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Heart valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 10 (10) | 18 (18)
Left ventricular dysfunction (Cardiac disorders) | 3 (3) | 2 (2)
Left ventricular failure (Cardiac disorders) | 11 (15) | 13 (13)
Mitral valve incompetence (Cardiac disorders) | 7 (8) | 6 (6)
Mitral valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 96 (104) | 108 (111)
Myocardial ischaemia (Cardiac disorders) | 47 (49) | 54 (61)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (3)
Pericarditis (Cardiac disorders) | 8 (12) | 4 (5)
Postinfarction angina (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 2 (2) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 2 (2)
Rheumatic heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 4 (4) | 4 (4)
Sinus arrest (Cardiac disorders) | 3 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 5 (5)
Sinus node dysfunction (Cardiac disorders) | 14 (14) | 13 (14)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 12 (12) | 6 (7)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 5 (6) | 5 (6)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 3 (3) | 1 (1)
Trifascicular block (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 2 (4)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 2 (2)
Ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 8 (8) | 9 (11)
Ventricular tachycardia (Cardiac disorders) | 19 (23) | 15 (21)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Congenital hepatobiliary anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diverticulitis meckel's (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Deafness neurosensory (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 11 (11) | 12 (13)
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 5 (5) | 8 (8)
Vestibular ataxia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 3 (3) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Adrenomegaly (Endocrine disorders) | 0 (0) | 2 (2)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 7 (7) | 8 (8)
Hyperadrenalism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1)
Amaurosis (Eye disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Amblyopia (Eye disorders) | 1 (1) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 28 (31) | 26 (32)
Cataract nuclear (Eye disorders) | 0 (0) | 2 (2)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1)
Corneal deposits (Eye disorders) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 3 (3) | 1 (1)
Diabetic retinopathy (Eye disorders) | 2 (2) | 2 (2)
Diplopia (Eye disorders) | 1 (1) | 3 (3)
Endocrine ophthalmopathy (Eye disorders) | 1 (1) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 2 (2)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Lagophthalmos (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 2 (2) | 0 (0)
Macular fibrosis (Eye disorders) | 2 (3) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Maculopathy (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 2 (4) | 4 (6)
Retinal haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Retinal vascular occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Tolosa-hunt syndrome (Eye disorders) | 0 (0) | 1 (1)
Tractional retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 4 (4) | 6 (7)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 4 (4) | 7 (7)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 9 (9)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 5 (7)
Acute haemorrhagic ulcerative colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 5 (5) | 11 (11)
Colitis ischaemic (Gastrointestinal disorders) | 7 (7) | 2 (2)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 13 (14) | 3 (3)
Diabetic gastroenteropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 11 (11)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 5 (6) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (5) | 2 (2)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (6) | 2 (2)
Enteritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 4 (4) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 9 (9) | 11 (11)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastritis (Gastrointestinal disorders) | 13 (15) | 20 (20)
Gastritis erosive (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 (18) | 18 (18)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 10 (10)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 3 (3)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Ileus (Gastrointestinal disorders) | 2 (3) | 4 (4)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 2 (2)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 10 (11) | 13 (13)
Intestinal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (4) | 4 (4)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 12 (12) | 9 (9)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Lumbar hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery embolism (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mesenteric panniculitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 (3) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palatal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 12 (12) | 12 (12)
Pancreatitis acute (Gastrointestinal disorders) | 13 (13) | 15 (17)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 10 (10) | 9 (9)
Small intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestine ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 5 (5) | 9 (10)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 8 (8)
Varices oesophageal (Gastrointestinal disorders) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 9 (9)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 4 (4) | 10 (10)
Cardiac death (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 29 (34) | 20 (20)
Complication associated with device (General disorders) | 1 (1) | 1 (1)
Critical illness (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 81 (81) | 89 (89)
Dehiscence (General disorders) | 1 (1) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 2 (2)
General physical health deterioration (General disorders) | 2 (2) | 5 (5)
Generalised oedema (General disorders) | 2 (2) | 0 (0)
Granuloma (General disorders) | 1 (1) | 1 (1)
Hernia (General disorders) | 2 (2) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 5 (5) | 3 (3)
Implant site inflammation (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 1 (1)
Inflammation (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 2 (2)
Medical device site irritation (General disorders) | 0 (0) | 1 (1)
Microlithiasis (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 9 (9) | 8 (8)
Necrobiosis (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 93 (110) | 107 (120)
Oedema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 5 (5)
Organ failure (General disorders) | 0 (0) | 1 (1)
Pacemaker syndrome (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pelvic mass (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 7 (14) | 13 (13)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0)
Stent-graft endoleak (General disorders) | 2 (2) | 0 (0)
Submandibular mass (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 14 (14) | 16 (16)
Sudden death (General disorders) | 21 (21) | 23 (23)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 2 (2)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 7 (8) | 8 (8)
Vascular stent thrombosis (General disorders) | 3 (3) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 9 (10) | 8 (8)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary dyspepsia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 11 (12) | 5 (6)
Cholangitis acute (Hepatobiliary disorders) | 4 (5) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 18 (18) | 22 (23)
Cholecystitis acute (Hepatobiliary disorders) | 25 (25) | 22 (22)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 6 (6)
Cholelithiasis (Hepatobiliary disorders) | 26 (26) | 38 (40)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 7 (8) | 11 (13)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 4 (4) | 3 (4)
Hepatic fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 4 (4)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Porcelain gallbladder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Allergy to metals (Immune system disorders) | 0 (0) | 1 (1)
Allergy to vaccine (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 2 (2)
Anaphylactic shock (Immune system disorders) | 3 (3) | 5 (5)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 3 (3)
Hashitoxicosis (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 2 (2)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 8 (8) | 9 (10)
Acquired immunodeficiency syndrome (Infections and infestations) | 1 (1) | 0 (0)
Acute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis b (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Amoebiasis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 5 (5) | 5 (5)
Appendiceal abscess (Infections and infestations) | 1 (3) | 1 (1)
Appendicitis (Infections and infestations) | 12 (12) | 12 (12)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 6 (6) | 11 (13)
Arthritis infective (Infections and infestations) | 1 (1) | 1 (1)
Aspergilloma (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 6 (6) | 3 (3)
Bacterascites (Infections and infestations) | 0 (0) | 1 (1)
Bacterial colitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bone abscess (Infections and infestations) | 1 (1) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 15 (16) | 35 (35)
Bronchitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 2 (2)
Burn infection (Infections and infestations) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 2 (2) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 84 (100) | 93 (117)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 6 (6) | 3 (3)
Chronic hepatitis c (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 7 (7) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 4 (5) | 1 (1)
Cystitis (Infections and infestations) | 9 (9) | 3 (3)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 3 (3)
Device related infection (Infections and infestations) | 4 (4) | 2 (2)
Diabetic foot infection (Infections and infestations) | 10 (11) | 13 (13)
Diabetic gangrene (Infections and infestations) | 7 (9) | 11 (11)
Diarrhoea infectious (Infections and infestations) | 3 (3) | 1 (1)
Diverticulitis (Infections and infestations) | 20 (24) | 20 (22)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 2 (2)
Encephalitis (Infections and infestations) | 3 (3) | 4 (4)
Encephalomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 4 (4) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 2 (2) | 2 (2)
Epiglottitis (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 11 (12) | 13 (13)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Escherichia sepsis (Infections and infestations) | 4 (4) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
External ear cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 2 (2) | 3 (4)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 22 (23) | 30 (40)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 26 (27) | 27 (27)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 5 (5)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 2 (2) | 2 (2)
H1n1 influenza (Infections and infestations) | 1 (1) | 1 (1)
Hiv infection (Infections and infestations) | 1 (1) | 1 (1)
Hiv-associated neurocognitive disorder (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 2 (2)
Helicobacter infection (Infections and infestations) | 1 (1) | 2 (2)
Hepatitis a (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis b (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 3 (3)
Human anaplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 4 (4) | 3 (3)
Infection (Infections and infestations) | 1 (1) | 6 (6)
Infectious colitis (Infections and infestations) | 3 (3) | 2 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 (4) | 1 (1)
Infective gastroduodenitis (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 17 (17) | 15 (15)
Intervertebral discitis (Infections and infestations) | 2 (2) | 4 (4)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Legionella infection (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 2 (2) | 4 (4)
Localised infection (Infections and infestations) | 16 (16) | 10 (11)
Lower respiratory tract infection (Infections and infestations) | 9 (11) | 10 (10)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Lyme disease (Infections and infestations) | 0 (0) | 2 (2)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 3 (3) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Medical device site abscess (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Medical device site joint infection (Infections and infestations) | 1 (1) | 2 (2)
Meningitis (Infections and infestations) | 1 (1) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (2) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Mucormycosis (Infections and infestations) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 2 (2) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 4 (4) | 5 (5)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 3 (3) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 3 (3)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 26 (35) | 39 (46)
Osteomyelitis acute (Infections and infestations) | 3 (3) | 3 (3)
Osteomyelitis chronic (Infections and infestations) | 4 (4) | 3 (3)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 3 (3)
Pelvic abscess (Infections and infestations) | 2 (3) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1) | 1 (1)
Perinephric abscess (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 5 (5)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pleurisy viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 194 (212) | 219 (246)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 5 (5)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 4 (4)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 9 (9) | 5 (5)
Postoperative abscess (Infections and infestations) | 3 (3) | 1 (1)
Postoperative wound infection (Infections and infestations) | 11 (11) | 13 (13)
Prostatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 3 (3)
Pyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 14 (14) | 14 (15)
Pyelonephritis acute (Infections and infestations) | 10 (10) | 15 (15)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 2 (2) | 3 (3)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 5 (7)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Rickettsiosis (Infections and infestations) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Salmonella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 4 (4)
Scrub typhus (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 77 (84) | 70 (71)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 21 (22) | 24 (27)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Splenic abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (2) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal infection (Infections and infestations) | 4 (4) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 5 (5)
Streptococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Tick-borne fever (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 2 (2) | 2 (2)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Urinary tract infection (Infections and infestations) | 49 (53) | 67 (71)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 22 (23) | 25 (26)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 5 (5) | 7 (8)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0)
Viral sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
West nile viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 11 (12) | 10 (11)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal wall wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 19 (19) | 14 (14)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 2 (4) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Cement embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Chest crushing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Costal cartilage fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 10 (10) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 14 (14) | 20 (20)
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 (5) | 9 (9)
Femur fracture (Injury, poisoning and procedural complications) | 16 (16) | 18 (18)
Fibula fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 4 (5) | 8 (8)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 13 (13) | 15 (16)
Humerus fracture (Injury, poisoning and procedural complications) | 11 (12) | 20 (20)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (4) | 3 (3)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 7 (8) | 4 (4)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 5 (5) | 9 (9)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Meniscus injury (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Patella fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 3 (5)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 8 (8) | 14 (14)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 11 (12) | 4 (5)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 7 (8) | 10 (10)
Rectal laceration postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 12 (13) | 15 (17)
Road traffic accident (Injury, poisoning and procedural complications) | 8 (8) | 7 (7)
Sedation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 12 (12) | 4 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 6 (6) | 9 (9)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 8 (9) | 11 (13)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 5 (5) | 8 (8)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Tibia fracture (Injury, poisoning and procedural complications) | 12 (12) | 5 (5)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 4 (4)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 2 (2)
Electrocardiogram st segment elevation (Investigations) | 1 (1) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 3 (3) | 0 (0)
Hepatitis c antibody positive (Investigations) | 0 (0) | 1 (2)
International normalised ratio increased (Investigations) | 0 (0) | 3 (3)
Liver function test increased (Investigations) | 2 (2) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Troponin i increased (Investigations) | 0 (0) | 1 (1)
Troponin t increased (Investigations) | 2 (4) | 0 (0)
Troponin increased (Investigations) | 11 (12) | 7 (8)
Urine cytology abnormal (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 20 (21) | 19 (19)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (6) | 13 (13)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 14 (14) | 29 (34)
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 27 (29) | 23 (27)
Diabetic ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 17 (23) | 27 (35)
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 3 (3) | 6 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 37 (49) | 55 (56)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (6) | 6 (7)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 69 (86) | 86 (101)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10) | 9 (9)
Hypovolaemia (Metabolism and nutrition disorders) | 14 (14) | 4 (4)
Ketoacidosis (Metabolism and nutrition disorders) | 7 (8) | 2 (2)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lipomatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 8 (8)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 7 (7) | 7 (7)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 14 (14) | 9 (9)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (9)
Bursitis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Immunoglobulin g4 related disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 24 (25) | 17 (18)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ligament calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 14 (15) | 18 (18)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle fibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 24 (25)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 103 (114) | 92 (102)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 16 (16)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 11 (11) | 12 (13)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (3)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 (20) | 18 (18)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 (42) | 27 (37)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 25 (25)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 8 (8)
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (3)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (20) | 20 (22)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (5)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7)
Chondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 6 (6)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 7 (7)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (17) | 16 (16)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Diffuse large b-cell lymphoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (8)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fallopian tube cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 8 (8)
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 4 (4)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 5 (5)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (7)
Lung adenocarcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 14 (14)
Lung carcinoma cell type unspecified stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (13) | 21 (21)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (17) | 12 (12)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 4 (4)
Malignant neoplasm of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant neoplasm of pleura metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 5 (7)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Non-hodgkin's lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 8 (8)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 9 (10)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Papillary tumour of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peritoneal carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 69 (70) | 55 (55)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostate cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 7 (8)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 8 (8)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Retro-orbital neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (12) | 10 (10)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (12)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 12 (14)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Vaginal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (2)
Arachnoid cyst (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 3 (3) | 1 (1)
Autonomic failure syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 1 (1)
Basilar artery perforation (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 3 (3) | 6 (6)
Brain oedema (Nervous system disorders) | 2 (2) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Brain stem infarction (Nervous system disorders) | 6 (8) | 3 (3)
Brain stem stroke (Nervous system disorders) | 2 (2) | 2 (2)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 5 (5) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 27 (27) | 21 (22)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 3 (3)
Cerebellar ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebellar infarction (Nervous system disorders) | 5 (5) | 2 (2)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 7 (7) | 6 (6)
Cerebral infarction (Nervous system disorders) | 24 (27) | 32 (33)
Cerebral ischaemia (Nervous system disorders) | 6 (6) | 9 (10)
Cerebrovascular accident (Nervous system disorders) | 102 (112) | 88 (94)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 3 (3) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 3 (4) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve palsies multiple (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 1 (1)
Dementia alzheimer's type (Nervous system disorders) | 3 (3) | 0 (0)
Dementia with lewy bodies (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 5 (5) | 4 (5)
Dizziness (Nervous system disorders) | 14 (14) | 9 (9)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 3 (3)
Dystonic tremor (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 2 (2) | 4 (4)
Encephalopathy (Nervous system disorders) | 3 (3) | 8 (8)
Epilepsy (Nervous system disorders) | 3 (3) | 5 (5)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 3 (3) | 8 (8)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 2 (3)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 3 (3)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 5 (5) | 11 (11)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 3 (4) | 4 (5)
Hydrocephalus (Nervous system disorders) | 2 (2) | 4 (4)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 2 (2)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Iiird nerve paralysis (Nervous system disorders) | 2 (2) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 97 (105) | 90 (99)
Lacunar infarction (Nervous system disorders) | 8 (9) | 14 (14)
Lacunar stroke (Nervous system disorders) | 2 (2) | 0 (0)
Lateral medullary syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 4 (4) | 6 (6)
Lumbar radiculopathy (Nervous system disorders) | 4 (4) | 6 (6)
Lumbosacral radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Medication overuse headache (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 4 (4) | 3 (3)
Migraine (Nervous system disorders) | 2 (2) | 2 (2)
Multiple system atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (2) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neurodegenerative disorder (Nervous system disorders) | 2 (2) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 2 (2) | 3 (6)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Postictal paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 3 (3)
Quadriplegia (Nervous system disorders) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 2 (2)
Radicular syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Radiculopathy (Nervous system disorders) | 2 (2) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 7 (7)
Seizure (Nervous system disorders) | 5 (6) | 10 (10)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Stiff person syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 37 (38) | 41 (44)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 2 (2) | 2 (2)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 2 (2) | 3 (3)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Toxic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 68 (76) | 54 (59)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vith nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Vith nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 2 (2)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 4 (4) | 5 (5)
Vertigo cns origin (Nervous system disorders) | 3 (3) | 2 (2)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Wernicke-korsakoff syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 3 (3) | 1 (1)
Device failure (Product Issues) | 0 (0) | 2 (2)
Device lead damage (Product Issues) | 2 (2) | 1 (1)
Device malfunction (Product Issues) | 3 (3) | 1 (2)
Device occlusion (Product Issues) | 2 (2) | 0 (0)
Stent malfunction (Product Issues) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 4 (4) | 12 (12)
Conversion disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 4 (4)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 13 (15)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 2 (2) | 6 (6)
Mental status changes (Psychiatric disorders) | 5 (5) | 7 (7)
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 2 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 1 (3)
Schizoaffective disorder depressive type (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 94 (96) | 127 (152)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 5 (5) | 6 (6)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 4 (4) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 9 (10) | 13 (17)
Cystitis glandularis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 2 (2) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis ulcerative (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 3 (3) | 2 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 3 (3) | 7 (8)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (4) | 16 (19)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 6 (6)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Myeloma cast nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 14 (16) | 18 (18)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 3 (3)
Oedematous kidney (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 5 (5)
Renal cyst (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 10 (11) | 17 (17)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (3) | 12 (12)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 3 (3)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)
Ureteric stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 5 (7) | 17 (21)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 5 (6)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary retention (Renal and urinary disorders) | 8 (8) | 10 (10)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 2 (2) | 5 (5)
Acquired phimosis (Reproductive system and breast disorders) | 11 (11) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 28 (30) | 31 (31)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hydrosalpinx (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile necrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 4 (4) | 8 (9)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 5 (5)
Rectocele (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Uterine prolapse (Reproductive system and breast disorders) | 6 (6) | 2 (2)
Uterovaginal prolapse (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Vaginal dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 37 (41) | 43 (50)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 18 (21)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 54 (81) | 54 (90)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 21 (22)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Paraneoplastic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 13 (14)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 10 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 27 (27)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (19)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 11 (11)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 15 (16)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 29 (30) | 24 (28)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 37 (45) | 29 (34)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Fixed eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 24 (28) | 23 (26)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 3 (3) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 12 (12) | 10 (11)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 22 (22) | 17 (17)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1)
Arterial insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Arterial perforation (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 4 (4) | 5 (5)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Arteritis (Vascular disorders) | 1 (2) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 3 (3)
Claudication of jaw muscles (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 17 (18) | 12 (12)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 3 (4) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2)
Essential hypertension (Vascular disorders) | 0 (0) | 3 (3)
Extremity necrosis (Vascular disorders) | 7 (7) | 4 (4)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery embolism (Vascular disorders) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 2 (2) | 6 (6)
Haemorrhagic vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 27 (28) | 27 (31)
Hypertensive crisis (Vascular disorders) | 14 (21) | 24 (28)
Hypertensive emergency (Vascular disorders) | 2 (2) | 7 (7)
Hypotension (Vascular disorders) | 28 (29) | 14 (14)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 2 (2)
Iliac artery disease (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 3 (3) | 2 (2)
Intermittent claudication (Vascular disorders) | 5 (5) | 3 (3)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 3 (3) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1)
Lymphatic fistula (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 6 (6) | 12 (13)
Peripheral arterial occlusive disease (Vascular disorders) | 43 (56) | 49 (53)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 14 (18) | 15 (20)
Peripheral artery stenosis (Vascular disorders) | 23 (36) | 20 (22)
Peripheral artery thrombosis (Vascular disorders) | 4 (5) | 4 (4)
Peripheral embolism (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 30 (32) | 35 (41)
Peripheral vascular disorder (Vascular disorders) | 34 (46) | 19 (21)
Peripheral venous disease (Vascular disorders) | 2 (2) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 2 (2) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava stenosis (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (2) | 2 (3)
Thromboangiitis obliterans (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 5 (6)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10 mg (N=8574) | Placebo (N=8569)
Acute kidney injury (Renal and urinary disorders) | 82 (91) | 112 (129)
Chronic kidney disease (Renal and urinary disorders) | 77 (78) | 104 (108)
Renal impairment (Renal and urinary disorders) | 121 (126) | 146 (159)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT01730534/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT01730534/SAP_001.pdf